CLINICAL TRIAL: NCT05501184
Title: COMPARISON OF SYNCHRONOUS AND ASYNCHRONOUS TELEREHABILITATION METHODS IN PATIENTS WITH CERVICAL DISC HERNIATION
Brief Title: SYNCHRONOUS AND ASYNCHRONOUS TELEREHABILITATION METHODS IN PATIENTS WITH CERVICAL DISC HERNIATION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Eren Timurtas, PhD, Marmara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26.05.2022/67
Record Dates: First submitted 2022-08-12; First posted 2022-08-15 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Cervical Disc Herniation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synchronous Telerehabilitation Group (Experimental): The exercise program was applied to groups that include three participants of the synchronous group 3 days per week by video conference method on an online platform (Zoom) with the supervision of a physiotherapist. The time of the group session was organized according to the availability of participants in that group and the physiotherapist using shared calendar availability (Doodle). The physiotherapist sent a reminder to participants one hour prior to each session including the video conference meeting link. Each exercise session lasted approximately 40 minutes. For 8 weeks, a total of 24 exercise sessions were performed. The physiotherapist demonstrated the exercises as needed, supervised the group by giving real-time feedback, and progressed the exercise program according to the needs of each group.
  Interventions: Other: Synchronous Exercise Program
- Asynchronous Telerehabilitation Group (Active Comparator): The exercise program was prescribed and followed up 3 days per week via the mobile application (FizyoTr). A notification was sent to participants' phones via mobile application prior to each session and attendance to the exercise program was recorded. For 8 weeks, a total of 24 exercise sessions were performed. The physiotherapist progressed the exercise program according to the assessment at 4 weeks and the needs of each participant.
  Interventions: Other: Asynchronous Exercise Program

INTERVENTIONS:
Other: Synchronous Exercise Program — The exercise program consisted of exercises by recommended guidelines for nonspecific neck pain patients which includes various strengthening, stretching, and proprioceptive exercises with progression.
  Arms: Synchronous Telerehabilitation Group
Other: Asynchronous Exercise Program — The exercise program consisted of exercises by recommended guidelines for nonspecific neck pain patients which includes various strengthening, stretching, and proprioceptive exercises with progression.
  Arms: Asynchronous Telerehabilitation Group

SUMMARY:
This was a randomized controlled trial conducted to examine the changes in the pain, physical function, quality of life, and kinesiophobia of participants with non-specific neck pain in Marmara University Physiotherapy and Rehabilitation Department. This study was approved by the Clinical Studies Ethics Committee of Marmara University Faculty of Health Sciences in January 2022 and was carried out in accordance with the Declaration of Helsinki. The participants were informed about the study and their consent was obtained.

ELIGIBILITY:
Inclusion Criteria:

* Participants between the ages of 18-65,
* Who had access to the internet and smartphone,
* Had the ability to conduct video calls were included in the study.

Exclusion Criteria:

* Participants were excluded if they had COVID-19,
* Had surgery in the last 6 months,
* Received physiotherapy treatment.
* Had a condition that prevented them from exercising.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating Scale (NPRS) | The pain was measured at baseline, mid-treatment in the 4th week, at the end of treatment in the 8th week, and a long-term follow-up assessment in the 16th week.
  Pain intensity was measured with a 0-10 cm scale. Participants were asked to rate their pain as "0: no pain and 10: excruciating pain" on the 0-10 cm scale (10). The pain reported by the patients was recorded in centimeters.

SECONDARY OUTCOMES:
Neck Disability Index (NDI) | The disability was measured at baseline, mid-treatment in the 4th week, at the end of treatment in the 8th week, and a long-term follow-up assessment in the 16th week.
  The participants' level of disability related to neck pain was evaluated using NDI. The NDI consists of 10 questions scored between 0 to 5 to measure disability related to limitation or pain (12). Questions include neck pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleep, and leisure activities. The scores range from 0 to 50 with higher scores indicating a more severe disability. The Turkish version of NDI has been shown to be valid and reliable in patients with neck pain
Tampa Scale of Kinesiophobia (TSK) | The kinesiophobia was measured at baseline, mid-treatment in the 4th week, at the end of treatment in the 8th week, and a long-term follow-up assessment in the 16th week.
  The TSK is a scale developed by Vlaeyen et al. consisting of 17 questions that assess kinesiophobia. For each question, a 4-point Likert scoring (1 = strongly disagree, 4 = completely agree) is used. After reversing items 4, 8, 12, and 16, a total score is calculated. The total score ranges from 17-68. A higher score indicates a higher level of kinesiophobia. The Turkish version of TSK has been shown to be valid and reliable.
Cervical Mobility | The cervical mobility was measured at baseline and at the end of treatment in the 8th week.
  The range of neck extension, flexion, and right and left lateral flexion were measured using a universal goniometer. For flexion and extension measurement, the participant sat on the side of the physiotherapist. The pivot point of the goniometer was placed at the acromion. The fixed arm of the goniometer was parallel to the ground. The measuring arm followed the midline of the ear. While measuring flexion, the participant was asked to try to touch his/her chin to the chest and for extension, to move his/her face parallel to the ceiling. For lateral flexion, pivot point of the goniometer was placed on the spinal ridge of C7. The fixed arm of the goniometer was kept parallel to the ground. The measuring arm followed the spinal projections of the vertebrae. The participant was asked to move his/her ear towards the shoulder.
Short Form-36 (SF-36) | The quality of life was measured at baseline and at the end of treatment in the 8th week.
  The quality of life was assessed using SF-36, which consists of 36 items. The Sf-36 has a total of 8 subscales including physical functioning, limitation due to physical problems (physical role), limitation due to emotional problems (emotional role), vitality, bodily pain, mental health, general health, and social functioning (19). The Turkish version of the SF-36 has been shown to have validity and reliability.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No